CLINICAL TRIAL: NCT04336306
Title: Cardiovascular Rehabilitation: Insertion of Virtual Reality-based Therapy and Evaluation of Barriers
Brief Title: Virtual Reality-based Therapy and Barriers in Cardiac Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mayara Moura Alves da Cruz, Principal Investigator, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29742920.9.0000.5402
Record Dates: First submitted 2020-03-31; First posted 2020-04-07 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Cardiovascular Diseases
Keywords: sympathetic nervous system; heart rate; blood pressure; virtual reality exposure therapy; barriers to cardiac rehabilitation; motivation; adherence patient; engagement; perceived exertion; oxygen saturation
MeSH Terms: conditions — Cardiovascular Diseases; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of chronic hemodynamic and autonomic repercussions (Experimental): Participants in a cardiovascular rehabilitation program will be randomly allocated to CR + VRBT interventions. This group will hold 3 weekly sessions (one for VRBT and two for CR) for 12 weeks. In the first, sixth and last week, chronic hemodynamic data and autonomic data will be evaluated.Furthermore,at the end of 12 weeks, a focus group with therapists and a focus group with patients will be held to identify qualitative aspects in relation to the insertion of VRBT. And in all eligible patients of CR wiil be applied the Questionnaire of barriers identification in frequenters of Cardiovascular Rehabilitation.
  Interventions: Other: virtual reality-based therapy (VRBT)

INTERVENTIONS:
Other: virtual reality-based therapy (VRBT) — The warm-up was performed using the "Just Dance 2015" game, in a sequence previously defined in a pilot study, aiming to increase HR progressively. A multimedia projector (Epson Power Life, H309A, China) connected to a console (Xbox One KinectTM, Microsoft, Redmond, WA) was used to project the game onto a white wall.The conditioning phase was performed using the "Shape Up" exercise game, in which patients perform exercises following a virtual therapist.

SUMMARY:
The aim of this study is to investigate the chronic hemodynamic and autonomic repercussions of the insertion of VRBT in CR. To qualitatively analyze the perception of patients and physiotherapists regarding the use of VRBT, as well as their association with CR, and through a new questionnaire that takes into account patients 'adherence, identifying which are the main barriers that influence patients' absences.

DETAILED DESCRIPTION:
Introduction: Despite the benefits that cardiovascular rehabilitation programs (CR) can promote, there are problems regarding adherence, which can be related to several factors, among them, motivation. Alternative therapies can reflect on motivation and promote increased adherence to CR. In this context, virtual reality-based therapy (VRBT) appears as an option. Additionally, chronic hemodynamic and autonomic repercussions of VRBT in relation to CV still need to be investigated. Objective: To evaluate the chronic hemodynamic and autonomic repercussions of the insertion of VRBT in CR. To qualitatively analyze the perception of patients and physiotherapists regarding the use of TRV, as well as their association with CR, and through a new questionnaire that takes into account patients 'adherence, identifying which are the main barriers that influence patients' absences. Methods: cardiac patients or individuals with factors that regularly participate in CR will participate in this study. Patients will be randomly allocated to CR + VRBT intervention or keeping the normal routine. Interventions will be carried out three times a week for 12 weeks. The primary outcome will be to assess chronic hemodynamic repercussions (blood pressure, heart rate, respiratory rate, oxygen saturation and perceived exertion using the Borg scale) and autonomic (linear and non-linear data). The secondary outcome consists of a qualitative assessment through a focus group with patients and a focus group with therapists, in addition, the new questionnaire developed to identify the influence of barriers on patients' adherence to CR will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cardiovascular disease.
* Clinical diagnosis of cardiovascular risk factors.

Exclusion Criteria:

* Presence exacerbated signs or symptoms.
* Balance problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2022-10-23 (Actual)

PRIMARY OUTCOMES:
Chronic autonomic response: linear indices | Change from baseline at 6 and 12 weeks
  Measured using heart rate variability : SDNN: the standard deviation of normal-to-normal intervals, ms; rMSSD: the root mean square of successive difference between normal intervals,ms; RRtri: triangular index, based on RR intervals,ms; TINN: triangular interpolation of the normal to normal interval between consecutive heart beats, ms; LF: low frequency, nu; HF: high frequency. In general higher values represent a better autonomic response.
Chronic autonomic response:no linear indices | Change from baseline at 6 and 12 weeks
  Measured using heart rate variability : Detrended Fluctuation Analysis, Recurrence Plot, Multiscalar Entropy, symbolic analysis.In general higher values represent a better autonomic response.
Blood pressure | Change from baseline at 6 and 12 weeks
  Measured using both systolic blood pressure and diastolic blood pressure
Heart rate | Change from baseline at 6 and 12 weeks
  Measured using an equipment validated for recording heart rate beat to beat
Respiratory rate | Change from baseline at 6 and 12 weeks
  Measured using the number of respiratory incursions in one minute
Oxygen Saturation | Change from baseline at 6 and 12 weeks
  Measured using an oximeter
Perceived Exertion | Change from baseline at 6 and 12 weeks
  Measured using Borg Scale, this scale varies from 6 to 20

SECONDARY OUTCOMES:
Perception of physiotherapists about the barriers and facilitators of the use of Virtual reality | After 12 weeks
  Measured by a focal groups with 5 therapist, that used virtual reality. Focal groups will be conducted by a researcher using a previously developed script, with open questions. The moderator will be a PhD student, with previous experience in physical training and qualitative research. A second researcher will be present at the focal groups to detail notes of the participant's answers.
Perception of patients about Virtual reality | After 12 weeks
  Measured by a 3 focal groups with 4 to 8 patients each, that performed virtual reality. Focal groups will be conducted by a researcher using a previously developed script, with open questions. The moderator will be a PhD student, with previous experience in physical training and qualitative research. A second researcher will be present at the focal groups to detail notes of the participant's answers.
Barriers identification in frequenters of Cardiovascular Rehabilitation. | After 12 week
  Measured by a new questionnaire of barriers. This new questionnaire has 15 questions, which are divided into domains.

CONTACTS AND LOCATIONS:
Overall Officials: Mayara MA da Cruz, Master, Principal Investigator — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- Universidade Estadual Paulista Júlio de Mesquita Filho, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alves da Cruz MM, Ricci-Vitor AL, Bonini Borges GL, Fernanda da Silva P, Ribeiro F, Marques Vanderlei LC. Acute Hemodynamic Effects of Virtual Reality-Based Therapy in Patients of Cardiovascular Rehabilitation: A Cluster Randomized Crossover Trial. Arch Phys Med Rehabil. 2020 Apr;101(4):642-649. doi: 10.1016/j.apmr.2019.12.006. Epub 2020 Jan 8. PMID 31926142
- [Background] da Cruz MMA, Ricci-Vitor AL, Borges GLB, da Silva PF, Turri-Silva N, Takahashi C, Grace SL, Vanderlei LCM. A Randomized, Controlled, Crossover Trial of Virtual Reality in Maintenance Cardiovascular Rehabilitation in a Low-Resource Setting: Impact on Adherence, Motivation, and Engagement. Phys Ther. 2021 May 4;101(5):pzab071. doi: 10.1093/ptj/pzab071. PMID 33625515
- [Result] da Cruz MMA, Grigoletto I, Ricci-Vitor AL, da Silva JM, Franco MR, Vanderlei LCM. Perceptions and preferences of patients with cardiac conditions to the inclusion of virtual reality-based therapy with conventional cardiovascular rehabilitation: A qualitative study. Braz J Phys Ther. 2022 May-Jun;26(3):100419. doi: 10.1016/j.bjpt.2022.100419. Epub 2022 May 18. PMID 35636061
- [Result] Alves da Cruz M, Laurino M, Christofaro D, Ghisi G, Vanderlei L. Long-term effects of virtual reality-based therapy in cardiovascular rehabilitation: A longitudinal study. Physiother Theory Pract. 2024 Apr;40(4):727-735. doi: 10.1080/09593985.2022.2160222. Epub 2022 Dec 25. PMID 36567613